CLINICAL TRIAL: NCT05776173
Title: Safety and Efficacy of Lentiviral Vector Transduction of β-globin Genetically Modified Autologous CD34+ Hematopoietic Stem Cells in Patients With Transfusion-dependent β-thalassemia
Brief Title: Safety and Efficacy of Gene Modified Autologous Hematopoietic Stem Cells to Treat Transfusion-dependent β-thalassemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai BDgene Co., Ltd. (Industry)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-TDT-211002
Record Dates: First submitted 2023-03-03; First posted 2023-03-20 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: β-thalassemia Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BD211 Single-Dose group (Experimental): Route of Administrate: infusion intravenously. Dosage form: injection solution. Dose: 5×10^6 cells /kg ~ 10×10^6 cells /kg. Frequency of administration: One dosing intravenously. Intervention: Single dose of BD211
  Interventions: Genetic: BD211

INTERVENTIONS:
Genetic: BD211 — Genetically modified CD34+ autologous stem cells were transfused intravenously with single dosing.

SUMMARY:
This study will be intented to evaluate the safety, tolerability, and engraftment efficacy after myeloablative preconditioning and transplantation of autologous CD34+ hematopoietic stem cells transduced with a lentiviral vector encoding the human βA-T87Q-globin gene in patients with transfusion-dependent (TDT) β-thalassemia.

DETAILED DESCRIPTION:
This is an open-label, single-dose study of BD211 in patients with transfusion-dependent β-thalassemia aged 6 to 35 years. It is estimated that 10 subjects will be enrolled. BD211 is a gene modified gene therapy product designed to produce healthy β-globin in red blood cells in beta-thalassemia patients. The total follow-up duration was 24 months, the safe endpoints and effectiveness endpoints will be used to assess the safety and efficacy profiles in patients with transfusion-dependent β-thalassemia.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 6 to 35 years old, including:

   Subjects should be able to provide an ICF. Diagnosed as Transfusion Dependent β-thalassemia with any genotype (β0, β+, βE/β0, βS/S, βS/β0, βS/β+), confirmed the Hb analysis. No alfa chain genetic abnormalities. Subjects must stabilize and maintain an appropriate iron chelation regimen. Transfusion-dependent types are defined as requiring at least 100 mL/kg/ year of red blood cells (pRBCs).
2. The tumor genes chip detection results about acute leukemia and myeloid tumor gene mutations (panel) showed no abnormality.
3. There were candidates for HLA gene semi-compatible hematopoietic stem cell transplantation.
4. No eligiblity for allogeneic hematopoietic stem cell transplantation.
5. The treatment of erythrocyte maturation agent luspatercept cannot be financially supported.
6. The investigator confirmed that subject was willing to follow the research procedures.
7. Having complete medical records including a history of blood transfusions testified subject received treatment and followed up for at least two years prior to screening.

Exclusion Criteria:

1. Availability of voluntary, fully HLA-matched hematopoietic cell donors, unless recommended for inclusion by the Monitoring Committee.
2. HIV-1 and HIV-2 were positive, and / or HTLV-1, HTLV-2 and VSV-G antibodies were positive.
3. An active bacterial, viral, fungal or parasitic infection.
4. Contraindicated for the extraction of bone marrow under anesthesia.
5. Any malignancy, myeloproliferative, or immunodeficient disease and relevant medical history.
6. Peripheral blood white blood cell (WBC) count < 3×10^9/L or platelet count < 120×10^9/L.
7. A history of allo-transplantation.
8. Erythropoietin was used within 3 months prior to HSC cell collection.
9. Immediate family members with known or suspected familial cancer syndromes (including but not limited to breast, colorectal, ovarian, prostate, and pancreatic cancers).
10. Subjects with a diagnosis of major mental illness may had a serious disability to participate in the study.
11. Active recurrent malaria.
12. Pregnant or postpartum nursing or unable to use contraception.
13. History of major organ injury including:

    Liver disease, transaminase > 3 times the upper limit of normal. (If the liver biopsy does not reveal evidence of widespread bridging fibrosis, cirrhosis, or acute hepatitis, this indicator will not be used as a criterion for the exclusion); Widely bridging fibrosis, histopathological evidence of acute hepatitis or cirrhosis showed in liver biopsy Heart disease, left ventricular ejection fraction < 25%; Kidney disease, creatinine clearance < 30% normal level; Of severe iron overload, confirmed by the study doctor; An heart MRI detection of T2 * < 10 ms; Significant pulmonary hypertension needing clinical medical intervention.
14. Any other conditions being ineligible for HSC transplantation determined by the investigator.
15. The subject involved with another clinical study in a 30-day screening period.
16. Subjects who expected to become parents during the 27-month study period.
17. Prior treatment with any type of gene and/or cell therapy.
18. As assessed by the investigator, the subjects or their parents are unable to comply well with the study procedures per protocol.
19. Hydroxyurea treatment within 3 months prior to hematopoietic stem cell collection.

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Red blood cell (RBCs) transfusion requirements, whether reaching TI | 24 months
  Comparison of blood volume and number of transfusions in the 2 years prior to participants enrolment as baseline with blood volume and number of transfusions up to months 6, 12, and 24 after receiving transfusion of the BD211.
  TI defined as peripheral blood weighted average hemoglobin (Hb) > or = 9 g/dL without pRBCs transfusion for 60 days after BD211 treatment, and transfusion is continuously halted for 12 months.
Total hospitalizing days at 6, 12, and 24 months (discharge after transplant) | 24 months
  Total hospitalizing days at 6, 12, and 24 months after transplantation were counted.

SECONDARY OUTCOMES:
Percentage of treated participants with Transfusion-Dependent β-Thalassemia (TDT) who achieved transfusion independence for at least 6 months | 24 months
  TI defined as peripheral blood weighted average hemoglobin (Hb) > or = 9 g/dL without pRBCs transfusion for 60 days after BD211 treatment, and transfusion is continuously halted for 12 months.
Change in RBCs infusion from baseline at 6 to 24 months | 24 months
  The quantity of RBCs transfusions at 6 to 24 months will be measured and compared with baseline level.
Mean Hb (g/dL) at 6, 12 and 24 months after treatment | 24 months
  Mean Hb (g/dL) in 6, 12, and 24 months after drug product infusion are tested and calculated.
Change in ferritin/liver iron levels from baseline | 24 months
  The Ferritin/liver iron levels are assayed per protocol plan, and evaluate the changes from those baseline level.
Neutrophil engraftment, platelet engraftment and vector copy number | 24 months
  Neutrophil engraftment was defined as the first of absolute neutrophil count (ANC) > or = 0.5 ×10^9/ L for 3 consecutive days (or 3 consecutive measurements done on separate days), after a post-transplant value less than (<) 0.5 × 10^9/L.
  Platelet engraftment was defined as the first of 3 consecutive platelet values > or =20 × 10^9/L for participants on different days with no platelet transfusionsadministered for 7 days immediately preceding. The day of engraftment is the first day of the 3 consecutive platelet measurements.
  Vector copy number will be detected per investigating time schedule.
Transplant-related mortality in 3 months and 12 months | 12 months
  Transplant related mortality was definedas any death occurring in the study post drug product infusion deemed related to the transplant bythe investigator.
Overall survival | 24 months
  Overall survival was defined as time from date of BD211 Drug Product infusion (Day 1) to date of death. Overall survival was censored at the date of last visit if the participant was still alive.
RCL incidence | 24 months
  Subjects blood RCL was detected with specific assay method, and the incidence was calculated at different scheduled timeslots.
Characterized insertion mutagenesis events that lead to clonal dominance or leukemia | 24 months
  The number of insertion mutagenesis events that characterized clonal dominance or leukemia was collected.
Frequency and severity of AE | 24 months
  An AE was any untoward medical occurrence associated with the use of a drug in participants, whether or not considered drug related. An AE may include a change in physical signs, symptoms, and/or clinically significant laboratory change occurring in any phase of a clinical study.

CONTACTS AND LOCATIONS:
Overall Officials: Sujiang Zhang, M.D., Principal Investigator — Ruijin Hospital, Shanghai, China
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No